CLINICAL TRIAL: NCT03710577
Title: Endocannabinoid and Psychological Responses to Yoga in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017-0980; A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW, Madison)
Record Dates: First submitted 2018-06-21; First posted 2018-10-18 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The proposed study is an acute, single group, crossover pilot study where participants will complete control and experimental conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): 40 minutes of Vinyasa yoga
  Interventions: Behavioral: Yoga
- Quiet Rest (Placebo Comparator): 40 minutes of quiet rest
  Interventions: Behavioral: Quiet Rest

INTERVENTIONS:
Behavioral: Yoga — 1 session
  Arms: Yoga
Behavioral: Quiet Rest — 1 session
  Arms: Quiet Rest

SUMMARY:
This study evaluates the acute effect of yoga on plasma levels of endocannabinoids and mood (i.e., mood disturbance, anxiety, pain) compared to one session of quiet rest. Participants completed one session of yoga and one session of quiet rest on two separate days.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years old and < 45 years old and
* report being healthy.

Exclusion Criteria:

* Being pregnant or planning to become pregnant,
* currently smoking,
* having a history of light headedness or fainting during blood draws or physical activity,
* having a history of chest pain during physical activity,
* having a bone, joint, cardiac, or other medical condition that a doctor has said may be worsened by physical activity,
* taking medications for any chronic diseases such as high blood pressure or diabetes,
* responding 'Yes' to any of the seven questions on the Par-Q.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Koltyn, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Natatorium, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited from students, faculty, and staff at the University of Wisconsin - Madison to participate in this study.
Pre-assignment Details: Volunteer eligibility was determined through a preliminary phone screen, participants were randomly assigned to receive the experimental task (Yoga) or the control task (quiet rest) first. Participants will then cross over 2-5 days after their first task to act as their own controls.
Groups:
- Yoga, Then Quiet Rest: 40 minutes of Vinyasa yoga Yoga: 1 session
  2-5 days between sessions
  40 minutes of quiet rest Quiet Rest: 1 session
- Quiet Rest, Then Yoga: 40 minutes of quiet rest Quiet Rest: 1 session
  2-5 days between sessions
  40 minutes of Yoga Yoga: 1 session
Period: First Intervention
Arm/Group | Yoga, Then Quiet Rest | Quiet Rest, Then Yoga
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Time Between Sessions (2-5 Days)
Arm/Group | Yoga, Then Quiet Rest | Quiet Rest, Then Yoga
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Yoga, Then Quiet Rest | Quiet Rest, Then Yoga
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Yoga, the Quiet Rest: 40 minutes of Vinyasa yoga Yoga: 1 session
  2-5 days between sessions
  40 minutes of Quiet Rest Quiet Rest: 1 session
- Total: Total of all reporting groups
Arm/Group | Yoga, the Quiet Rest | Quiet Rest, Then Yoga | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.75 (6.92) | 23 (3.16) | 24.83 (5.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants who marked their Ethnicity as 'Hispanic or Latino' also marked their Race as 'Hispanic or Latino'.
  Participants
    Race: American Indian or Native American | 0 | 0 | 0
    Race: Asian or Pacific Islander | 0 | 3 | 3
    Race: Black or African American | 0 | 0 | 0
    Race: White | 5 | 1 | 6
    Race: More than one race | 0 | 0 | 0
    Race: Hispanic or Latino | 3 | 0 | 3
    Race: Unknown or not reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Concentration of N-arachidonoylethanolamine
Description: Plasma concentration of anandamide, one effector of the endocannabinoid system
Time Frame: This will be measured 2 times during each study visit, once before the assigned study task (i.e., baseline) and once upon task completion (i.e., approx. 40 min. later)
Population: All participants for whom plasma samples were taken at baseline and post exercise
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Yoga | Quiet Rest
Number analyzed (Participants) | 9 | 8
pmol/mL | -.013 (.928) | -.655 (.724)

2. Primary Outcome: Change in Plasma Concentration of 2-Arachidonoylglycerol (2-AG)
Description: Plasma concentration of 2-AG, one effector of the endocannabinoid system
Time Frame: as for outcome 1
Population: All participants for whom plasma samples were taken at baseline and post exercise
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Yoga | Quiet Rest
Number analyzed (Participants) | 9 | 8
pmol/mL | .032 (.074) | -.008 (.049)

3. Secondary Outcome: Change in Total Mood Disturbance as Measured by the Profile of Mood States
Description: 65-item self-reported mood questionnaire that measures mood "right now." Scores range from 0-200 with higher scores indicating higher mood disturbance.
Time Frame: as for outcome 1
Population: All participants who completed the Profile of Mood States.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga | Quiet Rest
Number analyzed (Participants) | 12 | 12
score on a scale | -9.41 (9.12) | -7.17 (14.27)

4. Secondary Outcome: Change in State Anxiety as Measured by the State-Trait Anxiety Inventory
Description: 20-item self-reported anxiety questionnaire that measures anxiety "right now." Scores range from 20-80 with higher scores indicating higher anxiety.
Time Frame: as for outcome 1
Population: All participants who completed the State-Trait Anxiety Inventory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga | Quiet Rest
Number analyzed (Participants) | 12 | 12
score on a scale | -1.58 (10.48) | -1.92 (8.40)

5. Secondary Outcome: Change in Total Pain as Measured by the Short-form McGill Pain Questionnaire
Description: 15-item self-reported pain questionnaire that measures pain "right now." Scores range from 0-45 with higher scores indicating higher pain.
Time Frame: as for outcome 1
Population: All participants who completed the Short-form McGill Pain Questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga | Quiet Rest
Number analyzed (Participants) | 12 | 12
score on a scale | -1.50 (1.57) | 0.00 (2.63)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events while completing the research protocol on-site (i.e., 2 sessions on separate days, lasting about 1 hour each).
Arm/Group | Yoga | Quiet Rest
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03710577/Prot_SAP_000.pdf